CLINICAL TRIAL: NCT03474445
Title: Comparison of Two Volar Plating Systems for Distal Radius Fractures - A Prospective Randomized Single-blinded Controlled Clinical Trial
Brief Title: Comparison of Two Volar Plating Systems for Distal Radius Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Thomas Haider, Principal Investigator, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2339/2016
Record Dates: First submitted 2018-03-09; First posted 2018-03-22 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-04

CONDITIONS: Distal Radius Fracture
MeSH Terms: conditions — Wrist Fractures

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): Volar Plate Osteosynthesis Aptus 2.5
  Interventions: Procedure: Volar Plate Osteosynthesis Aptus 2.5
- Study Group (Active Comparator): Volar Plate Osteosynthesis Inteos 2.5
  Interventions: Procedure: Volar Plate Osteosynthesis Inteos 2.5

INTERVENTIONS:
Procedure: Volar Plate Osteosynthesis Aptus 2.5 — Volar plating of distal radius fracture. Device: Aptus 2.5
  Other Names: Henry approach, cutting of pronator quadratus
  Arms: Control group
Procedure: Volar Plate Osteosynthesis Inteos 2.5 — Volar plating of distal radius fracture. Device: Inteos 2.5
  Other Names: Henry approach, preservation of pronator quadratus
  Arms: Study Group

SUMMARY:
We plan to compare 2 types of plating systems for volar plating of distal radius fractures (Aptus 2.5® Medartis AG, Basel, Switzerland vs. INTEOS 2.5® - Hofer Medical GmbH and Co KG, Austria) in a prospective single-blinded controlled clinical trial.

DETAILED DESCRIPTION:
This study represents a prospective randomized clinical trial comparing two different systems of volar plate osteosynthesis in patients with distal radius fractures.

Patients meeting the inclusion criteria will be enrolled in the present study provided they give their consent. Informed written consent will be obtained. Envelopes will be prepared containing equal number of cards representing either the conventional or the novel plating syste. On the morning of the surgery a randomly picked envelope decides allocation one of the study groups. Patients will be blinded to treatment until completion of the study. Patients allocated to the control group receive Aptus 2.5® volar plate for distal radius fractures (Medartis AG, Basel, Switzerland), while patients in the study group will receive the plating system INTEOS 2.5® (Hofer GmbH and Co KG, Austria). In the control group, the pronator quadratus muscle will be cut prior mounting of the plate, while in the treatment group the plate will be inserted underneath the pronator quadratus leaving the muscle intact.

ELIGIBILITY:
Inclusion Criteria:

* " Distal radius fracture, Type A2, A3, B1, B2, B3, C1, C2 (according to AO Müller classification3) " Patient age between 18 and 75 years " Closed fracture or I° open fractures (according to Gustilo-Anderson classification6) " Agreement of patient to participate and written informed consent

Exclusion Criteria:

* " Polytraumatized patients " Severe systemic disorder (ASA 3) " New and/or preexisting fracture/Injury of contralateral forearm " II° and III° open fractures (according to Gustilo-Anderson classification6) " Associated injuries of the ipsilateral wrist (e.g. scapholunate dissociation, concomitant fractures) " Non-compliance to postoperative protocol (e.g. physiotherapy) " Delayed definitive surgical treatment of more than 14 days after injury " Change from temporary procedure (e.g. Fixateur externe) " Complex regional pain syndrome (CRPS, M.Sudeck) " Loss to follow-up

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Patient rated wrist evaluation | 12 months
  Outcome score based on a standardised questionnaire, 15 items, range 0-100, 0 =best possible score, 100=worst possible score

SECONDARY OUTCOMES:
Mayo wrist score | 8 weeks, 3 months, 6 months, 12 months
  Function-based evaluation of the wrist, range 0-100, 90-100=very good, 80-89=good, 65-79=satisfying, <65=poor
Radiological Outcome | 2weeks, 4 weeks, 8 weeks, 3 months, 6 months, 12 months
  x-ray based outcome of plate osteosynthesis (including ap and volar inclination angles, joint congruency, ulna length). Measurements will be performed on digitalised radiographs with IMPAX viewer (Agfa Ges.m.bH)
strength measurement | 4 weeks, 8 weeks, 3 months, 6 months, 12 months
  dynamometer-based strength evaluation
Volumetric evaluation | 4 weeks, 8 weeks, 3 months, 6 months, 12 months
  With a standardised device using water displacement wirst swelling will be assessed.
Disabilities of the Arm, Shoulder and Hand, Outcome Score - DASH | 4 weeks, 8 weeks, 3 months, 6 months, 12 months
  patient-based standardised questionnaire, 30 items, range 0-100, 0=best outcome, 100=worst outcome
Patient rated wrist evaluation | 4 weeks, 8 weeks, 3 months, 6 months
  Outcome score based on a standardised questionnaire, 15 items, range 0-100, 0 =best possible score, 100=worst possible score

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Haider, M.D., Ph.D., Principal Investigator — Medical University of Vienna
Locations (1):
- Medical Universtiy of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Thalhammer G, Hruby LA, Dangl T, Liebe J, Erhart J, Haider T. Does the pronator-sparing approach improve functional outcome, compared to a standard volar approach, in volar plating of distal radius fractures? A prospective, randomized controlled trial. J Orthop Traumatol. 2023 Apr 28;24(1):16. doi: 10.1186/s10195-023-00700-y. PMID 37118158